CLINICAL TRIAL: NCT00829985
Title: A Biomarker-based Pilot Study of Cockroach Sublingual Immunotherapy in Cockroach Sensitive Adults With Asthma and/or Perennial Allergic Rhinitis (ICAC-12)
Brief Title: Biomarker-based Cockroach Sublingual Immunotherapy Study (BioCSI)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Inner-City Asthma Consortium (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAIT ICAC-12; BioCSI (Other: NIAID)
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Results first posted 2013-03-08 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: Rhinitis, Allergic, Perennial; Asthma
Keywords: Rhinitis, Allergic, Perennial; Rhinitis, Allergic, Seasonal; Immunotherapy; Asthma; Nasal Allergies; Hypersensitivity
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Asthma; Rhinitis, Allergic, Seasonal; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glycerinated German Cockroach Allergenic Extract (Experimental): Participants with German cockroach allergy and mild to moderate asthma, rhinitis, or both self-administered concentrated (1:20 weight per volume [w/v]) daily doses of glycerinated German cockroach allergenic extract (50% glycerin) placed under the tongue (sublingually) to dissolve. The treatment course and study duration was 6 months. Note: The extract was also administered during the preliminary dosing visits, up to five escalating doses, or until the maximum study dose (420 microliters, 1:20 w/v) was achieved.
  Interventions: Biological: Glycerinated German Cockroach Allergenic Extract
- Placebo (Placebo Comparator): Participants with German cockroach allergy and mild to moderate asthma, rhinitis, or both self-administered daily doses of placebo placed under the tongue (sublingually) to dissolve. The treatment course and study duration was 6 months. Note: The placebo was also administered during the preliminary dosing visits, up to five escalating doses, or until the maximum study dose (420 microliters, 1:20 weight per volume [w/v]) was achieved.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Glycerinated German Cockroach Allergenic Extract — Concentrated (1:20 w/v) daily doses of glycerinated German cockroach allergenic extract placed under the tongue to dissolve. The extract is also administered during the preliminary dosing visits in up to five escalating doses or until the maximum study dose (420 microliters, 1:20 w/v) is achieved.
  Arms: Glycerinated German Cockroach Allergenic Extract
Biological: Placebo — Daily doses of cockroach allergenic extract placebo placed under the tongue to dissolve
  Arms: Placebo

SUMMARY:
There is currently no effective way to prevent development of allergic rhinitis (nasal allergies) and asthma and no cure. Sublingual immunotherapy (SLIT), a type of therapy in which allergens are placed under the tongue, may be a way to control and possibly prevent allergic rhinitis and asthma. However, detailed research of this approach is limited. The purpose of this study is to evaluate the safety and efficacy of a sublingual cockroach extract given to adults with perennial allergic rhinitis, asthma, or both.

DETAILED DESCRIPTION:
Over the last two decades, the prevalence of asthma has dramatically increased in many parts of the world. Currently, there are no effective ways to prevent the development of nasal allergies and asthma, and there are no cures for these diseases. Sublingual immunotherapy (SLIT) may help reduce symptoms of allergy and asthma. The purpose of this study is to evaluate the safety and efficacy of a cockroach extract given sublingually to adults with perennial (year-round) nasal allergies, asthma, or both.

At study entry, participants will receive a dose of placebo and then up to five incremental doses of cockroach extract or placebo at 15-minute intervals while observed by the clinical research staff. Doses will continue to be given until a sign or symptom occurs that indicates the participant is having difficulty tolerating the drug, or until the maximum study dose is reached.

For the next 6 months, participants will take the maximum study dose of cockroach extract or placebo daily at home.

This study will consist of 8 study visits. Skin tests, breathing tests, and blood collection will occur at study screening and other visits during the study. At study entry, participants will be taught to use an EpiPen in the event of a severe allergic reaction at any time during the study. A physical and oral exam, breathing test, and blood collection will occur at study entry and all follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* History of perennial allergic rhinitis, asthma, or both for a minimum of 1 year prior to study entry;
* Positive skin prick test to German cockroach;
* No known contraindications to therapy with glycerinated German cockroach allergenic extract or placebo; and
* Willing to sign the written Informed Consent prior to initiation of any study procedures.

Exclusion Criteria:

* Cannot perform spirometry at screening;
* Have clinically significant abnormal laboratory values;
* Have an Asthma classification of severe persistent at screening;
* Hospitalized for asthma within the 6 months prior to study entry;
* Life-threatening asthma exacerbation that required intubation, mechanical ventilation, or that resulted in a hypoxic seizure within the 2 years prior to study entry;
* No access to a telephone;
* Received allergen immunotherapy within the last 12 months prior to study entry and plan on initiating or resuming immunotherapy during the study;
* Treatment with anti-immunoglobulin E (anti-IgE) therapy within 1 year of study entry;
* Received an investigational drug within the 30 days prior to study entry and plan on using an investigational drug during the study;
* Experienced nausea, vomiting, abdominal pain or cramps, or diarrhea within the 3 months prior to study entry;
* Refuse to sign the Epinephrine Auto-injector Training Form;
* Does not primarily speak English;
* Plan to move from the area during the study period;
* History of idiopathic anaphylaxis or anaphylaxis grade 3;
* Using tricyclic antidepressants or beta-adrenergic blocker drugs;
* Clinically unacceptable complete blood count (CBC) and liver function tests, as defined by a hemoglobin less than 11.5 in males and 10.0 in females, or platelet counts less than 150,000 and an Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) greater than twice the upper limit of normal;
* Any condition that, in the opinion of the investigator, would interfere with the study; or
* Pregnant or breastfeeding.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wood, MD, Study Chair — Johns Hopkins University
Locations (4):
- United States (4):
  - National Jewish Center, Denver, Colorado
  - Childrens Memorial Hospital, Chicago, Illinois
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Boston University School of Medicine, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Participant level data and additional relevant materials are available to the public in the Immunology Database and Analysis Portal (ImmPort). ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.

REFERENCES:
- [Background] Ciprandi G, Contini P, Pistorio A, Murdaca G, Puppo F. Sublingual immunotherapy reduces soluble HLA-G and HLA-A,-B,-C serum levels in patients with allergic rhinitis. Int Immunopharmacol. 2009 Feb;9(2):253-7. doi: 10.1016/j.intimp.2008.11.009. Epub 2008 Dec 17. PMID 19100344
- [Background] Passalacqua G, Pawankar R, Baena-Cagnani CE, Canonica GW. Sublingual immunotherapy: where do we stand? Present and future. Curr Opin Allergy Clin Immunol. 2009 Feb;9(1):1-3. doi: 10.1097/ACI.0b013e3283196a9b. No abstract available. PMID 19106697
- [Background] Rolland JM, Gardner LM, O'Hehir RE. Allergen-related approaches to immunotherapy. Pharmacol Ther. 2009 Mar;121(3):273-84. doi: 10.1016/j.pharmthera.2008.11.007. Epub 2008 Dec 7. PMID 19111571
- [Result] Wood RA, Togias A, Wildfire J, Visness CM, Matsui EC, Gruchalla R, Hershey G, Liu AH, O'Connor GT, Pongracic JA, Zoratti E, Little F, Granada M, Kennedy S, Durham SR, Shamji MH, Busse WW. Development of cockroach immunotherapy by the Inner-City Asthma Consortium. J Allergy Clin Immunol. 2014 Mar;133(3):846-52.e6. doi: 10.1016/j.jaci.2013.08.047. Epub 2013 Nov 1. PMID 24184147
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) website — https://www.niaid.nih.gov/about/dait
- Available data/document: Individual Participant Data Set: SDY223 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY223 — ImmPort study identifier is SDY223.
- Available data/document: Study Protocol: SDY223 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY223 — ImmPort study identifier is SDY223.
- Available data/document: Study summary, -design, -adverse event(s), -interventions, -medications, -demographics, -study files.: SDY223 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY223 — ImmPort study identifier is SDY223.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Four National Institute of Allergy and Infectious Diseases (NIAID) Inner-City Asthma Consortium (ICAC) sites in the United States recruited the targeted number of study participants who fulfilled entry criteria between January and June 2009.
Period: Overall Study
Arm/Group | Glycerinated German Cockroach Allergenic Extract | Placebo
Started | 28 | 26
Completed | 19 | 22
Not Completed | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glycerinated German Cockroach Allergenic Extract | Placebo | Total
Number analyzed (Participants) | 28 | 26 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (9.9) | 33 (11.4) | 32 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 17 | 38
  Male | 7 | 9 | 16
Region of Enrollment [Number; unit: participants]
  United States | 28 | 26 | 54
German Cockroach-Specific Serum IgE Levels [Median (Full Range); unit: kU/L] | 1.9 [0.4 to 150] | 2.9 [0.4 to 113.3] | 2.0 [0.4 to 150]
German Cockroach-Specific Serum Immunoglobulin Subclass 4 (IgG4) Levels [Median (Full Range); unit: mg/mL] | 0.19 [0.01 to 3.59] | 0.08 [0.02 to 1.03] | 0.09 [0.01 to 3.59]

OUTCOME MEASURES:

1. Primary Outcome: Difference in German Cockroach-Specific Serum IgE Over Time
Description: Outcome is the ratio of geometric means for baseline German cockroach-specific serum Immunoglobulin E (IgE) vs. post-baseline German cockroach-specific serum IgE. This result is an indicator of immune modulation over time, however its clinical significance is unclear.
Time Frame: Baseline through 6-months of treatment
Population: Intent-to-treat
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Glycerinated German Cockroach Allergenic Extract | Placebo
Number analyzed (Participants) | 23 | 25
Ratio | 2.16 [1.81 to 2.57] | 1.12 [0.95 to 1.33]
Statistical Analysis 1: Comparison: Glycerinated German Cockroach Allergenic Extract vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Risk Ratio, log = 1.92, 95% CI 2-sided [1.51 to 2.45] — The estimated value and associated confidence interval represent the ratio of baseline-to-post-baseline change in the placebo group (denominator = 1.12) vs. the extract group (numerator = 2.16)

2. Secondary Outcome: Difference in German Cockroach-Specific Serum IgG4 Over Time
Description: Outcome is the ratio of geometric means for baseline German cockroach-specific serum Immunoglobulin subclass 4 (IgG4) vs. post-baseline German cockroach-specific serum IgG4. This ratio is an indicator of immune modulation, however its clinical significance is unclear.
Time Frame: Baseline through 6-months of treatment
Population: Intent-to-treat
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Glycerinated German Cockroach Allergenic Extract | Placebo
Number analyzed (Participants) | 23 | 25
Ratio | 1.06 [0.95 to 1.17] | 0.93 [0.83 to 1.03]
Statistical Analysis 1: Comparison: Glycerinated German Cockroach Allergenic Extract vs Placebo; Test type: Superiority or Other; p = 0.088, Mixed Models Analysis; Risk Ratio, log = 1.13, 95% CI 2-sided [0.98 to 1.32] — The estimated value and associated confidence interval represent the ratio of baseline-to-post-baseline change in the placebo group (denominator = 0.93) vs. the extract group (numerator = 1.06)

3. Secondary Outcome: Change in IgE Fragment Antibody Binding (FAB) Activity (30 Micrograms/mL Cockroach Allergen Extract)
Description: Outcome is the change in mean IgE fragment antibody binding (FAB) activity, baseline to post-baseline. Serum from sensitized donor incubated with 30 micrograms/mL of cockroach allergen extract in presence or absence of equal volume of sera from study participants to assess allergen-IgE binding. (Presence of sera from those who previously received allergen-specific immunotherapy, viz., study participants post-baseline, expected to inhibit allergen-IgE complex binding.) This change is an indicator of immune modulation, however its clinical significance is unclear.
Time Frame: Baseline through 6-months of treatment
Population: Intent-to-treat
Measure: Mean (95% Confidence Interval); unit: Percent antibody binding
Arm/Group | Glycerinated German Cockroach Allergenic Extract | Placebo
Number analyzed (Participants) | 23 | 25
Percent antibody binding | 4.7 [-1.72 to 11.28] | 0.7 [-5.56 to 6.87]
Statistical Analysis 1: Comparison: Glycerinated German Cockroach Allergenic Extract vs Placebo; Test type: Superiority or Other; p = 0.37, Mixed Models Analysis; Treatment Effect = 0.37, 95% CI 2-sided [-4.89 to 12.99] — Estimated value and associated confidence interval represent the treatment effect: change in the extract group (4.7) minus change in the placebo group (0.7)

4. Secondary Outcome: Change in IgE Fragment Antibody Binding (FAB) Activity (60 Micrograms/mL Cockroach Allergen Extract)
Description: Outcome is the change in mean IgE fragment antibody binding (FAB) activity, baseline to post-baseline. Serum from sensitized donor incubated with 60 micrograms/mL of cockroach allergen extract in presence or absence of equal volume of sera from study participants to assess allergen-IgE binding. (Presence of sera from those who previously received allergen-specific immunotherapy, viz., study participants post-baseline, expected to inhibit allergen-IgE complex binding.) This change is an indicator of immune modulation, however its clinical significance is unclear.
Time Frame: Baseline through 6-months of treatment
Population: Intent-to-treat
Measure: Mean (95% Confidence Interval); unit: Percent antibody binding
Arm/Group | Glycerinated German Cockroach Allergenic Extract | Placebo
Number analyzed (Participants) | 23 | 25
Percent antibody binding | 4.0 [-0.38 to 8.45] | -1.3 [-5.60 to 2.94]
Statistical Analysis 1: Comparison: Glycerinated German Cockroach Allergenic Extract vs Placebo; Test type: Superiority or Other; p = 0.09, Mixed Models Analysis; Treatment Effect = 5.4, 95% CI 2-sided [-0.77 to 11.51] — Estimated value and associated confidence interval represent the treatment effect: change in the extract group (4.0) minus change in the placebo group (-1.3)

5. Secondary Outcome: Percent of Participants With the Occurrence of Adverse Events (AE)
Description: Percent of participants who experienced at least one adverse event
Time Frame: Participant enrollment to end of study (up to 6 months post-baseline)
Population: Safety population
Measure: Number; unit: percentage of population
Arm/Group | Glycerinated German Cockroach Allergenic Extract | Placebo
Number analyzed (Participants) | 28 | 26
percentage of population | 93 | 85

ADVERSE EVENTS:
Arm/Group | Glycerinated German Cockroach Allergenic Extract | Placebo
Serious Adverse Events (participants affected / at risk) | 1/28 | 1/26
Other Adverse Events (participants affected / at risk) | 25/28 | 23/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glycerinated German Cockroach Allergenic Extract (N=28) | Placebo (N=26)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Scapula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glycerinated German Cockroach Allergenic Extract (N=28) | Placebo (N=26)
Ear pruritus (Ear and labyrinth disorders) | 7 (12) | 10 (11)
Eye pruritus (Eye disorders) | 5 (5) | 4 (4)
Lacrimation increased (Eye disorders) | 4 (5) | 3 (3)
Abdominal discomfort (Gastrointestinal disorders) | 2 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 7 (9) | 4 (9)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (9)
Oral mucosal erythema (Gastrointestinal disorders) | 2 (3) | 1 (1)
Oral pruritus (Gastrointestinal disorders) | 7 (18) | 8 (11)
Vomiting (Gastrointestinal disorders) | 4 (6) | 2 (2)
Adverse drug reaction (General disorders) | 9 (12) | 7 (9)
Chest discomfort (General disorders) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 2 (2)
Multiple allergies (Immune system disorders) | 2 (3) | 1 (2)
Seasonal allergy (Immune system disorders) | 2 (3) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Pharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 3 (4)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (5)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 12 (16) | 12 (21)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (9) | 8 (9)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (5)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No